CLINICAL TRIAL: NCT01598805
Title: Increased Rate of Prophylaxis Against Venous Thromboembolism Due to eAlerts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: FZMI-KEK-ZH-Nr. 2010-0458
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism/prevention & control
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- roll out of eAlerts (Experimental): Roll out of eAlerts providing evidence-based guidelines on prophylaxis against venous thromboembolism. An eAlert is displayed in the electronic patient chart if no prophylaxis has been ordered within 6 h after admission or transfer.
  Interventions: Behavioral: electronic alerts

INTERVENTIONS:
Behavioral: electronic alerts — An eAlert is displayed in the electronic patient chart if no prophylaxis has been ordered within 6 h after admission or transfer.
  Other Names: eAlert

SUMMARY:
Now, after a cluster randomized controlled trial, eAlerts providing evidence-based guidelines on venous thromboembolism prophylaxis will be rolled out and evaluated hospital-widely.

DETAILED DESCRIPTION:
An eAlert is displayed in the electronic patient chart if no prophylaxis has been ordered within 6 h after admission or transfer. The eAlerts provide evidence-based guidelines on venous thromboembolism prophylaxis. Now, after a cluster randomized controlled trial, the eAlerts will be rolled out and evaluated hospital-widely.

ELIGIBILITY:
Inclusion criteria:

* all in-patients hospitalized in a ward with computerized physician order entry (CPOE),
* staying at least 24 h in a ward

Exclusion criteria:

* outpatients,
* ward without CPOE,
* patients transferred from an intervention to a control ward and vice versa

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of prophylaxis against venous thromboembolism | 3 months
  patients with prophylaxis/total patients

SECONDARY OUTCOMES:
ordering time after admission or transfer of a patient | 3 months
  time when physicians order a venous thromboembolism prophylaxis
acceptance of the eAlerts | 3 months
  survey of compliant and incompliant physicians

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Blaser, Prof. PhD, Principal Investigator — University Hospital Zurich, Center for Clinical Research, Research Center for Medical Informatics
Locations (1):
- University Hospital Zurich, Center for Clinical Research, Zurich, Switzerland